CLINICAL TRIAL: NCT05388019
Title: Multidisciplinary Ventricular Assist Device Clinic: Feasibility Pilot Study and Quality of Life Impact Assessment
Brief Title: Multidisciplinary Ventricular Assist Device Clinic
Acronym: MultiVAD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Erin Coglianese, Medical Director, Mechanical Cardiac Support Program, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021P00351
Record Dates: First submitted 2022-05-11; First posted 2022-05-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Exercise Test

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prospective interventional cohort of newly-implanted patients (Experimental): This cohort will consist of patients who recently underwent LVAD implantation at Massachusetts General Hospital, and their caregivers. These patients will receive only multidisciplinary team care from the time of their implant.
  Interventions: Other: Multidisciplinary team clinic and assessments (Cardiopulmonary exercise test, six-minute-walk-test, MoCA, Quality of Life questionnaires)
- Prospective interventional cohort of previously-implanted patients (Experimental): This cohort will consist of patients who have previously undergone LVAD implantation at Massachusetts General Hospital who are being followed-up with standard-of-care VAD clinic visits, and their caregivers. These patients will receive a hybrid of multidisciplinary team care and standard-of-care visits.
  Interventions: Other: Multidisciplinary team clinic and assessments (Cardiopulmonary exercise test, six-minute-walk-test, MoCA, Quality of Life questionnaires)
- Retrospective control cohort (No Intervention): The historical control cohort will consist of retrospective data collection on patients who have undergone LVAD implantation in the past and no longer have an LVAD implanted (due to transplant, death, explant, etc.).
- Primary caregiver cohort (Experimental): This cohort will consist of primary caregivers of VAD patients from the two interventional cohorts. They will be administered a questionnaire at two timepoints. Each VAD patient will be associated with only one primary caregiver for the duration of the study.
  Interventions: Behavioral: Caregiver Self-Assessment

INTERVENTIONS:
Other: Multidisciplinary team clinic and assessments (Cardiopulmonary exercise test, six-minute-walk-test, MoCA, Quality of Life questionnaires) — Subject will receive care from a multidisciplinary team (physical therapy, occupational therapy, palliative care, social work) in addition to their standard of care VAD clinic visits. Subject will also perform a CPET, six-minute-walk-test, MoCA, and be administered quality of life questionnaires.
  Arms: Prospective interventional cohort of newly-implanted patients; Prospective interventional cohort of previously-implanted patients
Behavioral: Caregiver Self-Assessment — Primary caregivers of both interventional VAD patient cohorts will be administered a Caregiver Self-Assessment to assess burnout.
  Arms: Primary caregiver cohort

SUMMARY:
Current standard of care for ventricular-assist device (VAD) patients is composed of a multidisciplinary team (MDT), which is required in pre-implant and implant hospitalization care but is lacking in post-implant care. Post-implant care is currently centered around the avoidance of complications of VAD support, including cerebrovascular insult (CVA/TIA), gastrointestinal bleeding and infection. Despite major improvements in survival for VAD patients, quality of life and physical functioning measures have not seen significant improvements.

This study will include two prospective interventional cohorts and a retrospective control cohort. The first prospective interventional cohort will consist of patients who recently underwent LVAD implantation at Massachusetts General Hospital, and their caregivers. These patients will receive only multidisciplinary team care from the time of their implant. The second prospective interventional cohort will consist of patients who have previously undergone LVAD implantation at Massachusetts General Hospital who are being followed-up with standard-of-care VAD clinic visits, and their caregivers. These patients will receive a hybrid of multidisciplinary team care and standard-of-care visits. The historical control cohort will consist of retrospective data collection on patients who have undergone LVAD implantation in the past and no longer have an LVAD implanted (due to transplant, death, explant, etc.), and will be matched with the prospective interventional patients. The purpose of this study is to characterize the impact of routine MDT care on health-related quality of life, caregiver burnout and functional capacity of outpatient VAD patients, and to determine if implementation of MDT care is associated with a reduction in complications and readmissions in VAD patients at one- and two-years post implant. The investigators hypothesize that the MDT clinic model in addition to standard of care VAD management will positively impact the quality of life and functional status of VAD patients.

Subjects who consent to this study will be seen by the MDT providers and complete Cardiopulmonary Exercise Tests (CPET), six-minute-walk-tests, and quality of life questionnaires. The primary caregivers of these subjects will complete a Caregiver Self-Assessment at two timepoints. We anticipate to enroll 20 newly-implanted VAD patients in the pure-MDT arm, 35 pre-existing VAD patients in hybrid-MDT/SOC arm, and 55 primary caregivers.

DETAILED DESCRIPTION:
The current standard of care for ventricular-assist device (VAD) patients is composed of a multidisciplinary team (MDT), which is a mandated practice in the pre-implant and implant hospitalization phase of care. Each member of the MDT (surgeon, cardiologist, VAD coordinator, physical therapist, occupational therapist, social worker, and palliative care specialist) provides unique and orthogonal data. Post-implant care is currently centered around the avoidance of complications of VAD support, including cerebrovascular insult (CVA/TIA), gastrointestinal bleeding and infection. Although patients are referred to cardiac rehabilitation post VAD implant, assessment of functional capacity improvement post-implant is not well standardized. In our program, PT, OT, SW and palliative care medicine do not routinely see patients at intervals post-implant and are available in a limited fashion if specific concerns arise.

Prior studies have shown that MDT care in VAD patients improves survival in an in-patient setting and proves to be feasible and effective in other disease processes. Despite major improvements in survival for VAD patients however, quality of life and physical functioning measures have not seen significant improvements. Since there is a clinical need to examine post-implant treatment, this study aims to characterize the impact of routine MDT care on health-related quality of life, caregiver burnout and functional capacity of outpatient VAD patients, and to determine if implementation of MDT care is associated with a reduction in complications and readmissions in VAD patients at one- and two-years post implant.

This study will include two prospective interventional cohorts and a retrospective control cohort. The first prospective interventional cohort will consist of patients who recently underwent LVAD implantation at Massachusetts General Hospital, and their caregivers. These patients will receive only multidisciplinary team care from the time of their implant. The second prospective interventional cohort will consist of patients who have previously undergone LVAD implantation at Massachusetts General Hospital who are being followed-up with standard-of-care VAD clinic visits, and their caregivers. These patients will receive a hybrid of multidisciplinary team care and standard-of-care visits. The historical control cohort will consist of retrospective data collection on patients who have undergone LVAD implantation in the past and no longer have an LVAD implanted (due to transplant, death, explant, etc.). This group will be matched with the prospective interventional patients. The investigators hypothesize that the MDT clinic model in addition to standard of care VAD management will positively impact the quality of life and functional status of VAD patients. Future work will study readmission rates, medical complications, and overall survival difference between MultiVAD clinic care and usual care VAD clinics.

Subjects who consent to this study will be seen by the MDT providers and complete Cardiopulmonary Exercise Tests (CPET), six-minute-walk-tests, and quality of life questionnaires. Newly-implanted VAD subjects will participate over a 24-month period and previously-implanted VAD subjects will participate over a 12-month period. The primary caregivers of these subjects will complete a Caregiver Self-Assessment at two timepoints. We anticipate to enroll 20 newly-implanted VAD patients in the pure-MDT arm, 35 pre-existing VAD patients in hybrid-MDT/SOC arm, and 55 primary caregivers.

ELIGIBILITY:
Inclusion Criteria for Group A (newly-implanted):

* Ages 18+
* Individuals with ventricular assist device (VAD) implanted
* Individuals who have not previously attended standard-of-care VAD follow-up clinic visits

Exclusion Criteria for Group A:

* Inability to answer quality of life questionnaires
* Inability to perform the 6-minute walk test and Cardiopulmonary Exercise Test (CPET)
* Individuals who have previously attended standard-of-care VAD follow-up clinic visits

Inclusion Criteria for Group B (previously-implanted):

* Ages 18+
* Individuals with ventricular assist device (VAD) implanted
* Individuals who have previously attended standard-of-care VAD follow-up clinic visits

Exclusion Criteria for Group B:

* Inability to answer quality of life questionnaires
* Inability to perform the 6-minute walk test and CPET

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Peak VO2 in mL/kg of body weight/min during Cardiopulmonary Exercise Test | Change from pre-implant peak VO2 at 12 months post LVAD implantation
  Retrospective review in a patient chart.
Respiratory Exchange Ratio (RER) in % during Cardiopulmonary Exercise Test | Change from pre-implant RER at 12 months post LVAD implantation
  Retrospective review in a patient chart.
Minute ventilation per carbon dioxide production (VE/VCO2) during Cardiopulmonary Exercise Test | Change from pre-implant VE/VCO2 at 12 months post LVAD implantation
  Retrospective review in a patient chart.
Systolic and diastolic blood pressure in mmHg during Cardiopulmonary Exercise Test | Change from pre-implant blood pressure at 12 months post LVAD implantation
  Retrospective review in a patient chart.
Heart rate in beats per minute during Cardiopulmonary Exercise Test | Change from pre-implant heart rate at 12 months post LVAD implantation
  Retrospective review in a patient chart.
EuroQoL (EQ-5D and EuroVAS) to measure quality of life | Change from pre-implant up to 12 months post LVAD implantation
  Survey administered by research coordinator.
Kansas City Cardiomyopathy Questionnaire (KCCQ) to measure quality of life | Change from pre-implant up to 12 months post LVAD implantation
  Survey administered by research coordinator
Montreal Cognitive Assessment (MoCA) to measure cognitive function | Change from pre-implant up to 12 months post LVAD implantation
  Assessment administered by Occupational Therapist

SECONDARY OUTCOMES:
Number of readmissions | up to 24 months post-LVAD implantation
  Retrospective review in a patient chart
Time to readmission in days | up to 24 months post-LVAD implantation
  Retrospective review in a patient chart
Number of VAD related complications | up to 24 months post-LVAD implantation
  Retrospective review in a patient chart for GI bleed, CVA, heart failure, and infection

CONTACTS AND LOCATIONS:
Overall Officials: Erin Coglianese, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Tractenberg RE, Yumoto F, Aisen PS. Detecting When "Quality of Life" Has Been "Enhanced": Estimating Change in Quality of Life Ratings. Open J Philos. 2013 Nov 1;3(4A):24-31. doi: 10.4236/ojpp.2013.34A005. PMID 26213645